CLINICAL TRIAL: NCT01781559
Title: Effect of Phenolic Acids on the Human Vasculature
Brief Title: Bioefficacy of Phenolic Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11.35.NRC
Record Dates: First submitted 2013-01-28; First posted 2013-02-01 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — phenolic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- phenolic acid + maltodextrin (Experimental): phenolic acid + maltodextrin;
  Interventions: Dietary Supplement: phenolic acid
- Maltodextrin (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: phenolic acid
- flavanol + maltodextrin (Active Comparator): flavanol + maltodextrin
  Interventions: Dietary Supplement: phenolic acid

INTERVENTIONS:
Dietary Supplement: phenolic acid — phenolic acid

SUMMARY:
The objective is to demonstrate the effect of phenolic acids on endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Men and women
* Subjects with endothelial dysfunction defined as a basal brachial artery flow-mediated dilatation (FMD) measurement between 3% and 8% at screening

Exclusion Criteria:

* Any food allergy
* Abnormal blood pressure defined as follow: systolic <100 or >160 mmHg and diastolic <50 or >100mmHg
* Pregnancy or lactating women
* Regular consumption of cholesterol-lowering or antihypertensive medication
* Smokers
* Inability to restrain from caffeine/tea and alcohol for 12hrs prior to study visits (intake1 day before screening measurements (and 1 day before each visit)
* Not restrain the intake of multivitamin-tablets and other supplemental compounds 10 days before the study start and throughout the study.
* Excessive alcohol intake defined as > 280 g per week for men and >210g per week for women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from predose in percent change of flow-mediated dilatation at 1h compared to control treatment | After 1 hour

SECONDARY OUTCOMES:
Change from predose in blood pressure at 0.5h | After 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Croft, Professor, Principal Investigator — School of Medicine and Pharmacology - University of WA
Locations (1):
- School of Medicine and Pharmacology - University of WA, Perth, Australia